CLINICAL TRIAL: NCT03523546
Title: Oncology Episode Payment Model in Hawaii
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Hawaii Medical Service Association (Other)
Responsible Party: Principal Investigator, Amol Navathe, Principal Investigator, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 823981A
Record Dates: First submitted 2018-04-19; First posted 2018-05-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Colon Cancer; Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cancer Episode Payment Model (Experimental): Oncologists in this arm will be paid for each member's episode of care. The episode of care is 6 months in duration. Oncologists will have the opportunity to receive performance-based payments based upon a set of 6 quality metrics.
  Interventions: Other: Cancer Episode Payment Model (CEM)
- Fee for Service (No Intervention): Oncologists in this arm will not receive the intervention and will continue to be paid through fee-for-service.

INTERVENTIONS:
Other: Cancer Episode Payment Model (CEM) — Oncologists will be paid for an episode of care with the opportunity to receive a value based payment based on 6 quality metrics.
  Arms: Cancer Episode Payment Model

SUMMARY:
The HMSA Cancer Episode Payment Model (CEM) is a payment model designed to test the effects of better care coordination on health outcomes and costs of care for Hawaii Medical Services Association (HMSA) members with cancer who receive chemotherapy.

DETAILED DESCRIPTION:
The CEM is designed to improve community health, to improve care coordination, quality, and appropriateness of care, to improve patient experience, and to implement a value-based incentive structure that appropriately rewards oncologists for cost-savings and sustained of improved quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Any oncologist who practices with Hawaii Oncology and is a participating provider.

Exclusion Criteria:

* Any provider who does not practice with Hawaii Oncology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Composite quality score | 1 year
  Quality metrics included in the oncology model will be compared across the two arms.
Episode cost | 6 months
  Total spending of oncology patients in the episode will be compared across the two arms.
Utilization of acute and specialty care | 6 months
  Total utilization of acute and specialty care of oncology patients in the episode will be compared across the two arms

SECONDARY OUTCOMES:
Quality of care at end of life | 6 months
  Quality measures evaluating use of acute care and palliative care services at the end of life will be compared across the two arms
Survival | one year
  All cause mortality will be compared across the two arms

CONTACTS AND LOCATIONS:
Locations (1):
- Hawaii Oncology, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No